CLINICAL TRIAL: NCT00137956
Title: Endobronchial Valve for Emphysema PalliatioN Trial (VENT) Cost-effectiveness Sub-Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Emphasys Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 630-0005
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease
Keywords: Endobronchial Valve; Endobronchial Valve ProcedureEBV; EBV Procedure; Endobronchial Lung Volume Reduction; Lung Volume Reduction
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Device: Emphasys Endobronchial Valve (EBV) Device and Procedure

SUMMARY:
The purpose of the VENT Cost-Effectiveness Sub-Study is to gather healthcare utilization and quality of life information on patients enrolled in the VENT study in order to analyze the relative cost-effectiveness of the endobronchial valve implant procedure.

DETAILED DESCRIPTION:
Therapeutic interventions in health care require the use of resources. Since these resources are limited, it is important for clinical decision-makers to have economic information in addition to safety and efficacy data. In the economic environment of health care today, the incremental costs for a new therapeutic intervention must be offset by the value associated with better outcomes such as improved health and health-related quality of life and/or lower health care utilization costs over time.

Questions about the cost and effectiveness of medical care have generated considerable attention in medical outcomes research. In 1993, the Department of Health and Human Services appointed a multi-disciplinary group to recommend standards for the evaluation of health care. The panel's report suggested that standardized outcomes analyses be conducted to evaluate the cost-effectiveness of medical care. These analyses require preference-weighted measures of health-related quality of life. Such measures are needed in order to adjust survival time for health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by high-resolution computed tomography (HRCT) with eligible heterogeneous disease distribution
* Forced expiratory volume in 1 second (FEV1) < 45% predicted
* Total lung capacity (TLC) > 100% predicted
* Residual volume (RV) > 150% predicted
* Post rehabilitation 6 minute walk test > 140m
* Non-smoking for 4 months

Exclusion Criteria:

* Prior lung transplant, lung volume reduction surgery (LVRS), median sternotomy, bullectomy or lobectomy
* History of recurrent respiratory infections
* Evidence of large bullae (> 30% of either lung) in a non-target lobe
* FEV1 < 15% predicted
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 20% predicted

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2004-12

PRIMARY OUTCOMES:
The cost-effectiveness ratio in the treatment group as compared to the control group at 180 days

SECONDARY OUTCOMES:
The cost-effectiveness ratio in the treatment group of the study will be compared to established therapies and standards.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kaplan, PhD, Principal Investigator — UCLA School of Public Health, UCSD Health Outcomes Assessment Program (HOAP)

REFERENCES:
- [Background] Gold M, Franks P, Erickson P. Assessing the health of the nation. The predictive validity of a preference-based measure and self-rated health. Med Care. 1996 Feb;34(2):163-77. doi: 10.1097/00005650-199602000-00008. PMID 8632690
- [Background] Feeny D, Furlong W, Boyle M, Torrance GW. Multi-attribute health status classification systems. Health Utilities Index. Pharmacoeconomics. 1995 Jun;7(6):490-502. doi: 10.2165/00019053-199507060-00004. PMID 10155335
- [Background] Hays RD, Woolley JM. The concept of clinically meaningful difference in health-related quality-of-life research. How meaningful is it? Pharmacoeconomics. 2000 Nov;18(5):419-23. doi: 10.2165/00019053-200018050-00001. PMID 11151395
- [Background] Torrance GW, Furlong W, Feeny D, Boyle M. Multi-attribute preference functions. Health Utilities Index. Pharmacoeconomics. 1995 Jun;7(6):503-20. doi: 10.2165/00019053-199507060-00005. PMID 10155336
- [Background] Ware JE Jr, Gandek B. Overview of the SF-36 Health Survey and the International Quality of Life Assessment (IQOLA) Project. J Clin Epidemiol. 1998 Nov;51(11):903-12. doi: 10.1016/s0895-4356(98)00081-x. PMID 9817107
- [Background] Ramsey SD, Sullivan SD, Kaplan RM, Wood DE, Chiang YP, Wagner JL. Economic analysis of lung volume reduction surgery as part of the National Emphysema Treatment Trial. NETT Research Group. Ann Thorac Surg. 2001 Mar;71(3):995-1002. doi: 10.1016/s0003-4975(00)02283-9. PMID 11269488
- [Background] Ramsey SD, Berry K, Etzioni R, Kaplan RM, Sullivan SD, Wood DE; National Emphysema Treatment Trial Research Group. Cost effectiveness of lung-volume-reduction surgery for patients with severe emphysema. N Engl J Med. 2003 May 22;348(21):2092-102. doi: 10.1056/NEJMsa030448. Epub 2003 May 20. PMID 12759480
- [Background] Diabetes Prevention Program Research Group. Within-trial cost-effectiveness of lifestyle intervention or metformin for the primary prevention of type 2 diabetes. Diabetes Care. 2003 Sep;26(9):2518-23. doi: 10.2337/diacare.26.9.2518. PMID 12941712
- [Background] Kaplan RM. Value judgment in the Oregon Medicaid experiment. Med Care. 1994 Oct;32(10):975-88. doi: 10.1097/00005650-199410000-00001. PMID 7934274
- [Background] Sieber WJ, David KM, Adams JE, Kaplan RM, Ganiats TG. Assessing the impact of migraine on health-related quality of life: An additional use of the quality of well-being scale-self-administered. Headache. 2000 Sep;40(8):662-71. doi: 10.1046/j.1526-4610.2000.040008662.x. PMID 10971663
- [Background] Kaplan RM, Atkins CJ, Timms R. Validity of a quality of well-being scale as an outcome measure in chronic obstructive pulmonary disease. J Chronic Dis. 1984;37(2):85-95. doi: 10.1016/0021-9681(84)90050-x. PMID 6420431
- [Background] Kaplan RM, Anderson JP, Patterson TL, McCutchan JA, Weinrich JD, Heaton RK, Atkinson JH, Thal L, Chandler J, Grant I. Validity of the Quality of Well-Being Scale for persons with human immunodeficiency virus infection. HNRC Group. HIV Neurobehavioral Research Center. Psychosom Med. 1995 Mar-Apr;57(2):138-47. doi: 10.1097/00006842-199503000-00006. PMID 7792372
- [Background] Orenstein DM, Kaplan RM. Measuring the quality of well-being in cystic fibrosis and lung transplantation. The importance of the area under the curve. Chest. 1991 Oct;100(4):1016-8. doi: 10.1378/chest.100.4.1016. PMID 1914549
- [Background] Orenstein DM, Pattishall EN, Nixon PA, Ross EA, Kaplan RM. Quality of well-being before and after antibiotic treatment of pulmonary exacerbation in patients with cystic fibrosis. Chest. 1990 Nov;98(5):1081-4. doi: 10.1378/chest.98.5.1081. PMID 2225948
- [Background] Kaplan RM, Hartwell SL, Wilson DK, Wallace JP. Effects of diet and exercise interventions on control and quality of life in non-insulin-dependent diabetes mellitus. J Gen Intern Med. 1987 Jul-Aug;2(4):220-8. doi: 10.1007/BF02596443. PMID 3302144
- [Background] Ganiats TG, Palinkas LA, Kaplan RM. Comparison of Quality of Well-Being scale and Functional Status Index in patients with atrial fibrillation. Med Care. 1992 Oct;30(10):958-64. doi: 10.1097/00005650-199210000-00008. No abstract available. PMID 1405801
- [Background] Squier HC, Ries AL, Kaplan RM, Prewitt LM, Smith CM, Kriett JM, Jamieson SW. Quality of well-being predicts survival in lung transplantation candidates. Am J Respir Crit Care Med. 1995 Dec;152(6 Pt 1):2032-6. doi: 10.1164/ajrccm.152.6.8520772.
- [Background] Bombardier C, Ware J, Russell IJ, Larson M, Chalmers A, Read JL. Auranofin therapy and quality of life in patients with rheumatoid arthritis. Results of a multicenter trial. Am J Med. 1986 Oct;81(4):565-78. doi: 10.1016/0002-9343(86)90539-5. PMID 3532786
- [Background] Kaplan RM. Quality of life assessment for cost/utility studies in cancer. Cancer Treat Rev. 1993;19 Suppl A:85-96. doi: 10.1016/0305-7372(93)90061-u. PMID 7679324
- [Background] Kaplan RM. Decisions about prostate cancer screening in managed care. Curr Opin Oncol. 1997 Sep;9(5):480-6. doi: 10.1097/00001622-199709050-00014. PMID 9327227
- [Background] Patterson TL, Kaplan RM, Grant I, Semple SJ, Moscona S, Koch WL, Harris MJ, Jeste DV. Quality of well-being in late-life psychosis. Psychiatry Res. 1996 Jul 31;63(2-3):169-81. doi: 10.1016/0165-1781(96)02797-7. PMID 8878313
- [Background] Weinstein MC, Siegel JE, Gold MR, Kamlet MS, Russell LB. Recommendations of the Panel on Cost-effectiveness in Health and Medicine. JAMA. 1996 Oct 16;276(15):1253-8. PMID 8849754
- [Background] Russell LB, Gold MR, Siegel JE, Daniels N, Weinstein MC. The role of cost-effectiveness analysis in health and medicine. Panel on Cost-Effectiveness in Health and Medicine. JAMA. 1996 Oct 9;276(14):1172-7. PMID 8827972
- [Background] Weinstein MC, Stason WB. Foundations of cost-effectiveness analysis for health and medical practices. N Engl J Med. 1977 Mar 31;296(13):716-21. doi: 10.1056/NEJM197703312961304. PMID 402576
- [Background] Ries AL, Kaplan RM, Myers R, Prewitt LM. Maintenance after pulmonary rehabilitation in chronic lung disease: a randomized trial. Am J Respir Crit Care Med. 2003 Mar 15;167(6):880-8. doi: 10.1164/rccm.200204-318OC. Epub 2002 Dec 27. PMID 12505859